CLINICAL TRIAL: NCT02609906
Title: Operative Treatment of 2-fragment-fractures (AO 11-A3) of the Proximal Humerus in the Elderly: Cement Augmented Locking Plate Philos vs. Proximal Humerus Nail MultiLoc
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: LMU Klinikum (Other)
Responsible Party: Principal Investigator, Tobias Helfen, Dr. med. Tobias Helfen, LMU Klinikum
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 510-15
Record Dates: First submitted 2015-11-18; First posted 2015-11-20 (Estimated); Last update posted 2015-11-20 (Estimated); Status verified 2015-11

CONDITIONS: Shoulder Fractures; Intramedullary; Bone Plates
Keywords: proximal humerus; AO 11-A3 fracture; MultiLoc; Philos augmented
MeSH Terms: conditions — Shoulder Fractures

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PhilosTM with augmentation (Depuy-Synthes) (Other): The intervention group will be treated by the angle stable plate fixation system PhilosTM with augmentation (Depuy-Synthes)
  Interventions: Device: MultiLoc®-Nail (Depuy-Synthes)
- MultiLoc®-Nail (Depuy-Synthes) (Other): The comparison group will be treated by the multiplanar proximal humeral nail MultiLoc® (Depuy-Synthes).
  Interventions: Device: PhilosTM with augmentation (Depuy-Synthes)

INTERVENTIONS:
Device: PhilosTM with augmentation (Depuy-Synthes) — All fractures will initially be immobilised by a Gilchrist-bandage. This is the same procedure as for patients who do not attend this or any other trial and will be performed by the doctor on-duty in the emergency room. Patients will be admitted to the trauma ward after that. On the same day or at the latest on day after this patients will be informed about the current investigation, screened, included and randomized by one of the study doctors to our trial after written consent will be obtained as described above.
  Operative treatment is exclusively performed by the below mentioned study doctors. This group will be treated by the angle stable plate fixation system PhilosTM with augmentation (Depuy-Synthes).
  Arms: MultiLoc®-Nail (Depuy-Synthes)
Device: MultiLoc®-Nail (Depuy-Synthes) — All fractures will initially be immobilised by a Gilchrist-bandage. This is the same procedure as for patients who do not attend this or any other trial and will be performed by the doctor on-duty in the emergency room. Patients will be admitted to the trauma ward after that. On the same day or at the latest on day after this patients will be informed about the current investigation, screened, included and randomized by one of the study doctors to our trial after written consent will be obtained as described above.
  Operative treatment is exclusively performed by the below mentioned study doctors. This group will be treated by the multiplanar proximal humeral nail MultiLoc® (Depuy-Synthes).
  Arms: PhilosTM with augmentation (Depuy-Synthes)

SUMMARY:
Proximal humeral fractures are with an incidence of 4-5% the third most common fractures in the elderly. Compared to fractures of the upper limb it is the second most common fracture after distal radial fractures. 65% of all patients with a proximal humeral fracture are older than 60 years. Being aware of the demographic change there will even be an increase of incidence of these fractures. Kannus et al. showed an incidence of 298 per 100,000 in the at least 80 years old patients in 2007. Palvanen et al. predict an increase of incidence of 50% until 2030.

Approximately 80% of all humeral fractures are minimally or non-displaced and can be treated conservatively with a good functional result. In 20% of humeral fractures there is an indication for surgical treatment according to the modified Neer-Criteria. These criteria are fulfilled if there is an angulation of at least 45 degrees between fracture fragments, a displacement of the humeral shaft against the humeral head of at least 1 cm or a dislocation of the tuberculum of at least 5 mm.

Up to now there is evidence for superiority of any surgical treatment in literature. At the moment the most frequently used surgical technique for treatment of proximal humeral fractures is the angle stable plate fixation. There are various publications concerning this topic published by the investigators research group. In their 10-years results a majority of patients showed excellent and good, but also 16% showed unsatisfactory results after locking plate fixation. Main risk for poor outcome was revision surgery caused by secondary displacement (14%) which is also confirmed by results of other studies. In a further study investigators could show that there is a higher risk for secondary displacement in 2-part-fractures with a gross primary dislocation or a large metaphyseal fracture zone (AO 11-A3), especially in osteoporotic patients. More over these are common fractures and because of that a problem in surgical treatment.

A secondary varus dislocation of the head fragment and cutting-out are the most common complications of angle stable locking plates in AO 11-A3 fractures of the elderly. The primary reason for this mechanism of failure is certain instability of transmetaphyseal fractures in the region of the surgical neck caused by loss of impaction in a porous spongiosa. Because of that the forces on the head screws are high while the so called screw-bone-interface is rather weak after a surgical treatment.

Currently there exist various approaches to avoid a failure of the primary screw implantation. One possibility to increase the stability of the screw-bone-interface is the cement augmentation of the screw tips. To date there exist no clinical study that reports the results of locking plate fixation and the augmentation of cannulated head screws although it is a widely used method in everyday surgery, especially in the elderly.

A second possibility to prevent secondary displacement after surgical treatment of 2-fragment-fractures is the use of an intramedullary nails. A further development of intramedullary nails is multiplanar nailing. Screws can be inserted in various different levels and directions which can lead to a clearly higher stability.

A comparison of these two treatment options augmented locking plate versus multiplanar angle stable locking nail in 2-part proximal humeral fractures has not been carried out up to now.

DETAILED DESCRIPTION:
Because of the lack of clinical studies which compare cement augmented locking plates with multiplanar humeral nail systems after 2-part proximal humeral fractures, the decision of surgical method currently depends only on surgeons favour. Because only a randomized clinical trial (RCT) can sufficiently answer the question if one treatment option provides advantages compared to the other method we are planning to perform a RCT.

Investigators hypothesis: The cement augmented angle stable plate fixation system PhilosTM with augmentation (Depuy-Synthes) achieves significant differences concerning intra- and postoperative complication and revision rate, functional outcome and patient satisfaction compared to the multiplanar proximal MultiLoc®-Nail (Depuy-Synthes) in terms of Disabilities of the Shoulder, Arm and Hand-Score (DASH) Constant Score (CS), American Shoulder and Elbow Score (ASES), Oxford Shoulder Score (OSS), Range of motion (ROM) and Short Form 36 (SF-36).

ELIGIBILITY:
Inclusion Criteria:

* Age: ≤60 years or younger postmenopausal woman
* 2-fragment-fracture according to AO-classification AO 11-A3
* Signed informed consent
* Patient can read and understand German

Exclusion Criteria:

* Refusal to participate in the study
* Not Independent
* Dementia and/or institutionalized
* Does not understand written and spoken guidance German
* Pathologic fracture or a previous fracture of the same proximal humerus
* Alcoholism or drug addiction, e.g., in the emergency department, breathalyzer indicates blood alcohol concentration of more than 2%
* Other injury to the same upper limb requiring surgery
* Major nerve injury (e.g., complete radial- or axillary nerve palsy)
* Rotator cuff tear arthropathy
* Open fracture
* Multi-trauma or -fractured patient
* Fracture dislocation or head-splitting fracture
* Non-displaced fracture
* Isolated fracture of the major or minor tubercle
* Gross displacement of the fracture fragments (no bony contact between fracture parts or the humeral shaft is in contact with the articular surface)
* Any medical condition that excludes surgical treatment
* Pregnancy

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2015-11; Primary Completion 2016-11 (Estimated)

PRIMARY OUTCOMES:
Disabilities of the Shoulder, Arm and Hand-Score (DASH) | 24 months
  Funcitonal outcome

SECONDARY OUTCOMES:
Constant Score (CS) | 24 months
  Funcitonal outcome
American Shoulder and Elbow Score (ASES) | 24 months
  Funcitonal outcome
Oxford Shoulder Score (OSS) | 24 months
  Funcitonal outcome
Range of motion (ROM) | 24 months
  Funcitonal outcome
Short Form 36 (SF-36) | 24 months
  Life quality
Barthel Index | 24 months
  Life quality

CONTACTS AND LOCATIONS:
Locations (1):
- Munich University Hospital, Munich, Bavaria, Germany

REFERENCES:
- [Result] Kannus P, Palvanen M, Niemi S, Sievanen H, Parkkari J. Rate of proximal humeral fractures in older Finnish women between 1970 and 2007. Bone. 2009 Apr;44(4):656-9. doi: 10.1016/j.bone.2008.12.007. Epub 2008 Dec 24. PMID 19135560
- [Result] Palvanen M, Kannus P, Niemi S, Parkkari J. Update in the epidemiology of proximal humeral fractures. Clin Orthop Relat Res. 2006 Jan;442:87-92. doi: 10.1097/01.blo.0000194672.79634.78. PMID 16394745
- [Result] Neer CS 2nd. Displaced proximal humeral fractures. I. Classification and evaluation. J Bone Joint Surg Am. 1970 Sep;52(6):1077-89. No abstract available. PMID 5455339
- [Derived] Handoll HH, Elliott J, Thillemann TM, Aluko P, Brorson S. Interventions for treating proximal humeral fractures in adults. Cochrane Database Syst Rev. 2022 Jun 21;6(6):CD000434. doi: 10.1002/14651858.CD000434.pub5. PMID 35727196
- [Derived] Helfen T, Siebenburger G, Mayer M, Bocker W, Ockert B, Haasters F. Operative treatment of 2-part surgical neck fractures of the proximal humerus (AO 11-A3) in the elderly: Cement augmented locking plate Philos vs. proximal humerus nail MultiLoc(R). BMC Musculoskelet Disord. 2016 Oct 28;17(1):448. doi: 10.1186/s12891-016-1302-6. PMID 27793135